CLINICAL TRIAL: NCT07181434
Title: Impact of Virtual Reality on Patient Pain During Lower Limb Revascularization Via Endovascular Surgery Under Local Anesthesia With Sedation - Randomized Study
Brief Title: Impact of Virtual Reality on Patient Pain During Lower Limb Revascularization Via Endovascular Surgery Under Local Anesthesia With Sedation
Acronym: REVDOU
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: REVDOU
Record Dates: First submitted 2025-08-08; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Peripheral Arterial Disease
Keywords: Virtual reality; pain management; virtual reality headset
MeSH Terms: conditions — Peripheral Arterial Disease; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In addition to the usual care, the patient will be equipped with VR headsets (Experimental): In addition to the usual care, the patient will be equipped with VR headsets showing one of the six scenes from the HealthyMind® program in 3D, accompanied by hypnotic speech during the procedure.
  Interventions: Device: The patient will be equipped with VR headsets
- The patient will receive the usual treatment under local anesthesia (No Intervention): The patient will receive standard care under local anesthesia with an analgesic injection (paracetamol) +/- morphine sedation (remifentanil), according to the treatment protocol and tailored to the patient.

INTERVENTIONS:
Device: The patient will be equipped with VR headsets — The patient will be equipped with VR headsets showing one of the six scenes from the HealthyMind® program in 3D, accompanied by hypnotic speech during the procedure.
  Arms: In addition to the usual care, the patient will be equipped with VR headsets

SUMMARY:
The prevalence of peripheral arterial disease (PAD) increases with age In addition to medical treatment, endovascular procedures can be performed, depending on the stage of the disease, to prevent complications and/or sequelae (relapse, functional loss of the affected limb, amputation, death), but also to relieve pain. This is a minimally invasive procedure most often performed under local anesthesia (LA), sometimes with the administration of sedatives (morphine and analgesics) to relieve pain and reduce anxiety related to the procedure.

Non-pharmacological methods such as virtual reality (VR) are increasingly being used as an alternative to general anesthesia and excessive opioid use.

The hypothesis is that VR could reduce pain during lower limb revascularization by endovascular surgery.

DETAILED DESCRIPTION:
The prevalence of peripheral arterial disease (PAD) increases with age. In high-income countries, it is 5% between the ages of 45 and 49, and 18% after the age of 85. In France, nearly 1 million people are affected by this disease.

In addition to medical treatment, endovascular procedures can be performed, depending on the stage of the disease, to prevent complications and/or sequelae (relapse, functional loss of the affected limb, amputation, death), but also to relieve pain. This is a minimally invasive procedure most often performed under local anesthesia (LA), sometimes with the administration of sedatives (morphine and analgesics) to relieve pain and reduce anxiety related to the procedure.

Local anesthesia causes discomfort related to the operating environment (low temperature, harsh lighting, noise, supine position, arms along the body, cold, hard, narrow table), impacting patient cooperation and making the procedure difficult, with the need to take multiple X-rays and reinject potentially nephrotoxic contrast agents. It can lead to the procedure being stopped, with serious consequences (postponement, persistent or even worsening pain, amputation, death).

Non-pharmacological methods such as virtual reality (VR) are increasingly being used as an alternative to general anesthesia and excessive opioid use.

It has proven effective in managing pain and anxiety during various medical, surgical, and endovascular procedures. Its high-quality graphics immerse the patient; hypnotic speech and relaxing elements capture the patient's attention; breathing exercises help manage stress; and relaxing music creates a soothing atmosphere. This support ensures greater mental and physical comfort by reducing pain and anxiety.

The hypothesis is that VR could reduce pain during lower limb revascularization by endovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient suffering from PAD, scheduled to undergo endovascular surgery for lower limb revascularization under local anesthesia combined with sedation.
* Age ≥ 18 years.
* Patient who understands and speaks French.
* Patient covered by social security or covered through a third party.
* Free subject, without guardianship, curatorship, or subordination.
* Patient who has given their free and informed consent.

Exclusion Criteria:

* Patients with contraindications to VR headsets (mono- or binocular blindness, epilepsy, migraines, psychiatric disorders, pacemakers, hearing aids, defibrillators, recent injuries to the eyes, face, or scalp that prevent comfortable use of the headsets, etc.).
* Patients with suspected intolerance to VR headsets (sensitivity to motion sickness in cars, history of balance or eye disorders, etc.);
* Previous bad experience with VR headsets;
* Patients undergoing local regional anesthesia (LRA);
* Persons requiring enhanced protection, namely persons deprived of their liberty by judicial or administrative decision, pregnant women, and finally patients in life-threatening situations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
The maximum intensity of pain experienced by the patient during the procedure will be measured at the end of the procedure using the numerical pain scale (EN) ranging from 0 for "no pain" to 10 for "worst pain imaginable." | At the end of the revascularization procedure of the lower limbs by endovascular surgery

SECONDARY OUTCOMES:
Anxiety will be measured at Baseline and just after the intervention using an EN ranging from 0 for "no anxiety" to 10 for "maximum imagined anxiety" | At Baseline and just after the intervention of lower limb revascularization through endovascular surgery
  Anxiety will be measured at Baseline and just after the intervention using an EN ranging from 0 for "no anxiety" to 10 for "maximum imagined anxiety": a quick, easy-to-use scale that correlates strongly with Spielberger's STAI scale (Benotsch et al., 2000).
Systolic Blood Pressure (SBP) in mmHg | At Baseline before the procedure of lower limb revascularization through endovascular surgery, upon arrival in the operating room, then every 15 minutes until the end of the procedure.
Diastolic Blood Pressure (DBP) in mmHg | At Baseline before the procedure of lower limb revascularization through endovascular surgery, upon arrival in the operating room, then every 15 minutes until the end of the procedure.
Heart Rate (HR) in cycles/min | At Baseline before the procedure of lower limb revascularization through endovascular surgery, upon arrival in the operating room, then every 15 minutes until the end of the procedure.
Respiratory Rate (RR) in Beats Per Minute (BPM) | At Baseline before the procedure of lower limb revascularization through endovascular surgery, upon arrival in the operating room, then every 15 minutes until the end of the procedure.
Total doses and classes of analgesics, morphine derivatives, and anesthetics consumed | During the procedure of lower limb revascularization through endovascular surgery
The dose of X-ray radiation | During the procedure of revascularization of the lower limbs by endovascular surgery
  Total dose of X-ray radiation absorbed by the patient (dose-area product, in mGy.cm²)
The volume of contrast medium delivered | During the procedure of revascularization of the lower limbs by endovascular surgery
The difference between the duration of the procedure as perceived by the patient and the actual duration of the procedure in minutes | At the end of the procedure of revascularization of the lower limbs by endovascular surgery
The success rate of the procedure | At the end of the procedure of revascularization of the lower limbs by endovascular surgery
  Proportion of procedures performed successfully (total revascularization of the artery)
Proportion of patients who kept the virtual reality headsets on throughout the procedure | Throughout the procedure of lower limb revascularization through endovascular surgery
VR satisfaction score, rated on a scale from 0 for "not at all satisfied" to 10 for "completely satisfied." | At the end of the procedure of lower limb revascularization through endovascular surgery

CONTACTS AND LOCATIONS:
Locations (1):
- C.H.U. Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No